CLINICAL TRIAL: NCT05015621
Title: A Phase 3, Randomized, Open-label, Multi-center Study to Evaluate the Efficacy and Safety of Surufatinib Plus Toripalimab Versus FOLFIRI as a Secondline Treatment in Patients With Advanced Neuroendocrine Carcinoma
Brief Title: A Phase 3 Study to Evaluate Surufatinib Plus Toripalimab in the Treatment of Advanced Neuroendocrine Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-012-00CH1
Record Dates: First submitted 2021-08-08; First posted 2021-08-20 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Advanced Neuroendocrine Carcinoma
Keywords: secondline treatment in patients
MeSH Terms: interventions — surufatinib; toripalimab; Fluorouracil; Leucovorin; Irinotecan; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): all subjects will receive study treatment in 21-day cycle, Surufatinib 250mg, QD and Toripalimab, 240mg, IV drip, Q3W, D1, the treatment will continue until one of the following conditions occurs: progression of disease, death, intolerable toxicity, or the end of study treatment (as other criteria specified in the protocol are met), whichever occurs first
  Interventions: Drug: Surufatinib plus Toripalimab
- control group (Other): FOLFIRI group subjects will receive study treatment in 14- day cycle, Irinotecan: 180 mg/m^2, iv drip over 30～90 minutes, on Day 1; Calcium folinate: 400 mg/m^2, iv drip for about 2 hours, given upon completion of infusion of Irinotecan on Day 1; 5-FU: 400 mg/m^2, iv bolus, given upon completion of infusion of Calcium folinate on Day 1, followed by 2400 mg/m^2 continuously iv drip for 46～48 hours.
  Interventions: Drug: 5-fluorouracil, Calcium folinate and Irinotecan

INTERVENTIONS:
Drug: Surufatinib plus Toripalimab — Surufatinib is a tablet in the form of 50mg, oral, once a day; Toripalimab is an injection in the form of 240mg, intravenous, once three weeks.
  Other Names: HMPL-012 plus JS001
  Arms: study group
Drug: 5-fluorouracil, Calcium folinate and Irinotecan — Irinotecan 180 mg/m^2, Calcium folinate 400 mg/m^2, 5-FU total 2800 mg/m^2 will be administrated once two weeks.
  Other Names: FOLFIRI
  Arms: control group

SUMMARY:
To evaluate the efficacy of Surufatnib combined with Toripalimab compared with FOLFIRI in the treatment of advanced neuroendocrine carcinoma

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, multicenter, phase III clinical study designed to evaluate the efficacy and safety of surufatnib combined with toripalimab compared with FOLFIRI in patients with advanced neuroendocrine carcinoma who have progression of disease or intolerable toxicity after previous 1st-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who included in this study must fulfil all of the following criteria:

  1. Fully aware of this study and voluntary to sign the informed consent form (the informed consent form must be signed before any trial-specific procedure is performed);
  2. Aged 18~75 years (inclusive);
  3. Histologically or cytologically confirmed, unresectable, locally advanced or metastatic neuroendocrine carcinoma
  4. Patients with neuroendocrine carcinoma who have failed previous platinum-based 1st-line chemotherapy
  5. ECOG performance status of 0 or 1 ;
  6. Having clear measurable lesions as defined by RECIST v1.1;
  7. Patients who agree to provide tumor specimens for pathological type review and biomarkers detection;
  8. Patients with adequate bone marrow, liver and kidney organ functions whose laboratory tests within 7 days before the first dose meet the following requirements:

     1. Absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥100×109/L and hemoglobin ≥90 g/dL (without blood transfusion or use of blood products for correction within 14 days prior to laboratory examination, and without use of granulocyte colony stimulating factor or other hematopoietic stimulating factor for correction within 7 days prior to laboratory examination);
     2. Serum total bilirubin ≤1.5 × upper limit of normal (ULN);
     3. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤2.5 × ULN in the absence of liver metastases; ALT and AST ≤5 × ULN in the presence of liver metastases.
     4. Serum creatinine ≤ 1.5 × ULN and creatinine clearance ≥ 50 mL/min (calculated according to the Cockcroft-Gault formula, see Appendix 3);
     5. Routine urinalysis showing urine protein < 2+; in case of urine protein ≥ 2+, 24-hour urine protein (quantitative) should be <1g;
     6. International normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (APTT) ≤1.5 × ULN.
  9. Estimated survival ≥ 12 weeks;
  10. Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose. Male or female patients of childbearing potential volunteer to use effective contraceptive methods during the study and within 90 days after last administration of the study drug, such as double barrier contraception, condoms, oral or injectable contraceptives, intrauterine contraceptive device, etc. All female patients will be considered to be of childbearing potential unless they are naturally postmenopausal, underwent artificial menopause, or are surgically sterile (e.g., hysterectomy, bilateral adnexectomy).

Exclusion Criteria:

* Subjects must be excluded from this study when any one of the following criteria is met:

  1. Toxicities associated with previous anti-tumor treatment do not return to ≤CTCAE grade 1, except for alopecia and peripheral neurotoxicity (≤ CTCAE grade 2 ) caused by Oxaliplatin;
  2. Presence of other malignancies in the past 5 years (except for basal cell carcinoma or squamous cell carcinoma of the skin and carcinoma in situ of the cervix, which were effectively controlled);
  3. Presence of central nervous system (CNS) metastases in screening period;
  4. Use of approved systematic anti-tumor therapy within 4 weeks prior to the first dose, including chemotherapy, biotherapy, targeted therapy (the washout period of small molecular targeted drugs lasts 2 weeks or 5 half-lives, whichever is shorter), hormone therapy, treatments with traditional Chinese medicine (for patients receiving treatments with traditional Chinese medicine with clear anti-tumor indications, for anti-tumor indications clearly specified in the package insert, one-week washout period prior to the first dose is acceptable), etc.;
  5. Use of radical radiotherapy (including radiotherapy for more than 25% of the bone marrow) within 4 weeks before the first dose; brachytherapy (e.g. radioactive particle implantation) within 60 days prior to the first dose; palliative radiotherapy for bone metastases within 1 week before the first dose;
  6. Previous use of anti (PD-1), anti-PD-L1, anti-PD-L2 or CTLA-4 antibody or any other antibody acting on T cell co-stimulatory or checkpoint pathways
  7. Previous use of vascular endothelial growth factor (VEGF)/vascular endothelial growth factor receptor (VEGFR) targeted therapy;
  8. Previous therapy with Irinotecan;
  9. Having abnormal thyroid function with symptoms ongoing or requiring treatment at screening ;
  10. Use of immunosuppressant within 4 weeks prior to the first dose, not including local glucocorticoid via nasal spray, inhalation or other routes or systemic glucocorticoid at physiological dose (i.e., no more than 10mg/day of prednisone or equivalent dose), temporary use of glucocorticoid for treatment of dyspnea resulted from asthma, chronic obstructive pulmonary disease is allowed, and preventive use of corticosteroid to avoid allergic reactions is allowed
  11. Patients with any active autoimmune disorders requiring systematic treatment or a history of autoimmune disease in the past 2 years,
  12. Use of systemic immune stimulants within 4 weeks prior to the first dose;
  13. Vaccination of any live or attenuated live vaccine within 4 weeks prior to the first dose or during the study.
  14. Patients having received major surgical operation within 4 weeks prior to the first dose .
  15. Uncontrollable malignant hydrothorax, ascites or pericardial effusion ;
  16. Patients who currently have hypertension that cannot be controlled by medication.
  17. Patients who currently have any disease or condition that affects drug absorption, or patient who cannot take the drug orally;
  18. Use of CYP3A potent or moderate inducers during the administration of concomitant medications or within 2 weeks or 5 half-lives (whichever is longer) prior to the first dose;
  19. Patients who currently have gastric and duodenal active ulcer, ulcerative colitis, or active bleeding in the unresected tumor, or serious gastrointestinal disorders , or other conditions that may cause haemorrhage of digestive tract or perforation
  20. Patients with evidence or history of obvious bleeding tendency within 2 months prior to the first dose
  21. Arterial thrombosis or deep venous thrombosis occurred within 6 months prior to the first dose; or stroke events and/or transient ischemic attacks occurred within 12 months.
  22. Clinically significant cardiovascular disorder,
  23. Presence of clinically significant electrolyte abnormality judged by the investigator;
  24. Patients with active infection or fever of unknown origin during screening and prior to the first dose (body temperature >38.5°C);
  25. Patients with active tuberculosis (TB), receiving anti-tuberculosis therapy currently or within one year prior to the first dose;
  26. Patients with pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, serious lung function impairment that may interfere with the detection and management of suspected drug-related pulmonary toxicities; radiation pneumonitis in the area of radiotherapy is allowed;
  27. Human immunodeficiency virus (HIV) antibody positive;
  28. Patients with known history of clinically significant liver diseases, including those infected with active viral hepatitis [HBV DNA > 1 × 104 copies/mL or > 2000 IU/mL when hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HbcAb) is positive; patients with known positive hepatitis C virus antibody (HCV Ab) and HCV RNA > 1 × 103 copies/mL], or other hepatitis, including moderate and severe hepatic cirrhosis with a clinical significance;
  29. Use of clinical drug treatment which has not been approved or marketed in China within 4 weeks prior to the first dose;
  30. Pregnant (positive pregnancy test prior to administration) or lactating women;
  31. Patients with known allergy to any component of toripalimab, surufatnib or Irinotecan, fluorouracil and calcium folinate preparations, or previous history of serious allergy to any other monoclonal antibody;
  32. Patients with other reasons that, in the opinion of the investigator, make it unsuitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2021-09-18 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of first dose of study drug until withdrawal of consent or death (up to approximately 2 years)
  Duration from the date of initial treatment to the date of death due to any cause.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) (RECIST1.1) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anticancer therapy (up to approximately 2 years)
  A duration from the date of initial treatment to disease progression or death of any cause.
Objective response rate (ORR)(RECIST1.1) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anticancer therapy(up to approximately 2 years)]
  The incidence of confirmed complete response or partial response
Duration of response (DoR)(RECIST1.1) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anti-cancer therapy (up to approximately 2 years)]
  Duration from the first time reported partial response or complete response to the first time of disease progression or death.
Disease control rate (DCR)(RECIST1.1) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anti-cancer therapy (up to approximately 2 years)]
  Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit.
PD-L1 | Baseline (before the randomization)
  To evaluate the relationship between the efficacy and tumor biomarkers of PD-L1
Ki67 | Baseline (before the randomization)
  To evaluate the relationship between the efficacy and tumor biomarkers of ki67
Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) | From the within 7 days prior to the initiation of treatment to 30 days after the last administration
  The changes in health-related quality of life (HRQoL) score from baseline and the time to deterioration of symptoms (TTD) as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Prof., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No